CLINICAL TRIAL: NCT07005388
Title: CULTURAL ADAPTATION OF GROUP CBT PSYCHOSIS MANUAL AND ESTABLISHING ITS EFFICACY IN PAKISTAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Punjab Institute of Mental Health (Other Government)
Responsible Party: Principal Investigator, Nazish Habib, Clinical Psychologist, Punjab Institute of Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIMHclinicalTrials
Record Dates: First submitted 2024-03-21; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Psychotic Disorders; Psychosis; Schizophrenia and Related Disorders
Keywords: Group CBT; CBT; schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive behavioral therapy for psychosis (Experimental): Experimental group given CBTp
  Interventions: Behavioral: Cognitive behavioral therapy for psychosis

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for psychosis — Cognitive behavioral therapy for psychosis is a group protocol design specially for psychotic patients to treat their positive and negative symptoms

SUMMARY:
A study aimed to culturally adapt group Cognitive Behavioral Therapy for psychosis (CBTp) for Pakistani patients with schizophrenia. Fifty inpatients from PIMH were randomly assigned to experimental (N=25) and control (N=25) groups. Both groups showed significant improvement in symptoms post-intervention (p<0.05). This suggests that culturally adapted group CBTp is effective for schizophrenia patients in hospital settings, addressing the scarcity of CBT-trained therapists in government hospitals in Pakistan.

DETAILED DESCRIPTION:
A clinical trial was conducted aiming to culturally adapt and pilot test a group Cognitive Behavioral Therapy for psychosis (CBTp) protocol for Pakistani patients diagnosed with schizophrenia spectrum disorder. This research was particularly significant given the prevalence of psychosis in Pakistan and the scarcity of trained therapists, especially in government hospitals.

Methodology:

Participant Selection: Purposive sampling was utilized to select participants from the Psychiatric Institute of Mental Health (PIMH) who were diagnosed with schizophrenia spectrum disorder and were inpatients receiving medication.

Sample Size: A total sample of N=50 was obtained, with participants randomly assigned to either the experimental (N=25) or control group (N=25).

Assessment Measures: Various assessment measures were employed to evaluate the efficacy of the intervention, including the Positive and Negative Syndrome Scale of Schizophrenia (PANSS), Rosenberg's Self Esteem Scale, Insight Scale, Brief COPE, Perceived Stress Scale, and The Psychotic Symptom Rating Scales (PSYRATS).

Intervention: The experimental group received manualized group CBT intervention consisting of 24 sessions over a duration of 3 months. The intervention was culturally adapted to suit the needs and context of Pakistani patients. Importantly, there were no dropouts from either group during the intervention period.

Statistical Analysis: An analysis of covariance (ANCOVA) was conducted to compare pre- and post-intervention ratings between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

A clinical diagnosis of schizophrenia or psychotic disorder for at least 5 years.

Aged between 18 and 65.

The exclusion criteria :

A severe learning disability, an organic brain disorder , a high level of disturbed behavior, or a significant risk of suicide or homicide.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
PANSS and self esteem scale | 6
  Different scales according to treatment protocol were used

CONTACTS AND LOCATIONS:
Locations (1):
- Punjab Institute of mental health, Lahore, Punjab Province, Pakistan